CLINICAL TRIAL: NCT02119897
Title: Feasibility Study Evaluating Extraorally Delivered Low Level Light Therapy (LLLT) for the Prevention of Oropharyngeal Mucositis in Pediatric Patients Undergoing Myeloablative Hematopoietic Cell Transplantation
Brief Title: Feasibility Study of Low Level Light Therapy for Prevention of Oropharyngeal Mucositis in Pediatric Transplants Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nathaniel S. Treister, DMD, DMSc, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 13-611
Record Dates: First submitted 2014-04-09; First posted 2014-04-22 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Oropharyngeal Mucositis; Myeloablative Hematopoietic Cell Transplantation; Low Level Light Therapy
Keywords: Oropharyngeal Mucositis; Myeloablative Hematopoietic Cell Transplantation; Low Level Light Therapy
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low Level Light Therapy (LLLT) (Experimental): * LLLT: The LLLT device will be positioned next to the face and neck for a total of 6 exposures: Right face, Midline face, Left face, Left neck, Midline neck, Right neck
  * Dose per anatomic site 50mW/cm2, 60 sec = 3.0J/cm2
  * Route: Extraoral
  * Total Treatment Time (all sites): 6 min
  * Schedule: Participants will be treated daily (including weekends and holidays) beginning on the first day of HCT conditioning and continuing through day +20 or hospital discharge if prior to day +20.
  * Evaluation: Participants will undergo formal mucositis and toxicity assessments at baseline and daily from day -1 through day +20, with a final assessment on the last day of treatment.
  Interventions: Device: Low Level Light Therapy

INTERVENTIONS:
Device: Low Level Light Therapy
  Other Names: THOR Model LX2M (THOR Photomedicine Ltd, Chesham, UK)

SUMMARY:
Oral mucositis (OM) is a painful and potentially debilitating acute toxicity that frequently affects children undergoing hematopoietic cell transplantation (HCT). As a result of intensive conditioning with chemotherapy with or without total body irradiation, and in the case of allogeneic HCT, graft-versus-host disease (GVHD) prophylaxis, patients are at risk for developing diffuse ulcerations of the oral and esophageal mucosa that result in pain and suffering, increased utilization of opioid analgesics, and the need for intravenous or total parenteral nutritional support. Patients universally report OM as being the worst aspect of the HCT experience.A novel approach has been the use of larger light-emitting diode arrays to treat the at risk tissues from an extraoral approach, enabling exposure of the oral, oropharyngeal, and esophageal mucosa while avoiding the need for intraoral manipulation, and requiring only minimal patient cooperation. In this research study, the investigators are assessing the feasibility of providing extraorally delivered low level light therapy (LLLT) for the prevention of OM in children undergoing myeloablative HCT.

DETAILED DESCRIPTION:
This is an open label, single treatment arm clinical pilot study. The study is targeted to enroll twelve evaluable patients

OBJECTIVES:

Primary

* Determine the feasibility of providing extraoral LLLT for prevention of OM in pediatric patients undergoing HCT

Secondary

* Determine the feasibility of collecting data using the WHO Oral Toxicity Scale and ChIMES in pediatric patients undergoing myeloablative HCT who are treated with extraoral LLLT for prevention of OM
* Evaluate the safety and tolerability of extraoral LLLT for prevention of OM in pediatric patients undergoing myeloablative HCT

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo myeloablative conditioning followed by autologous or allogeneic hematopoietic cell transplantation at Boston Children's Hospital.
* 4 years of age to 25 years of age.
* WHO Oral Toxicity score of 0 at baseline evaluation (first day of conditioning).
* Ability to understand and the willingness to sign a written informed consent document (for patients under the age of 18 this applies to parent/guardian)
* Ability to understand and/or the willingness of their parent or legally authorized representative to sign a written informed consent document.

Exclusion Criteria:

* Treatment with oral LLLT within 4 weeks of HCT.
* Participants may not be receiving any other agents intended for the prevention/management of mucositis (including palifermin and ice chips/cryotherapy).
* WHO ≥1 at baseline evaluation.

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The ability to maneuver and provide a new treatment for mucositis using (extraoral) LLLT | 20 Days
  Several measures will be collected to evaluate the overall feasibility of providing daily extraoral LLLT for children undergoing HSCT including:
  * Accessibility and maneuverability of the LLLT device (transportation from storage site to hospital room, device weight)
  * Administration of LLLT (device settings, positioning of device, delivery of therapy)
  * Patient tolerability (level of comfort during treatments, compliance with daily therapy
  * Proportion of days with therapy administered, as evidence by data submitted (goal is ≥75%)
  * Ability to enroll at least 5 patients within the first 3 months (this pertains to the feasibility of study conduct, and not to the feasibility of the therapeutic approach)

SECONDARY OUTCOMES:
Patient compliance with completing questionnaires | 2 Years
  To address secondary the investigators, will calculate the following proportion: (number of times patients refused to complete one or both questionnaires) / (number of questionnaire completion timepoints), and place a 95% confidence interval on the proportion.
WHO Oral Toxicity Scale/ChIMES Instrument | 2 Years
  To address secondary aim, the investigator, will analyze the data from the WHO Oral Toxicity Scale and the ChIMES instrument using the analytic methods specifically prescribed for these standardized instruments.
Toxicity measured using CTC Version | 2 Years
Dose-limiting toxicity | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Treister, DMD,DMSc, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Treister NS, London WB, Guo D, Malsch M, Verrill K, Brewer J, Margossian S, Duncan C. A Feasibility Study Evaluating Extraoral Photobiomodulation Therapy for Prevention of Mucositis in Pediatric Hematopoietic Cell Transplantation. Photomed Laser Surg. 2016 Apr;34(4):178-84. doi: 10.1089/pho.2015.4021. Epub 2016 Mar 16. PMID 26982624